CLINICAL TRIAL: NCT02417961
Title: A Multicenter, Open-Label, Functionality, Reliability, and Performance Study of an Accessorized Pre-filled Syringe With Home-administered Subcutaneous Benralizumab in Adult Patients With Severe Asthma (GREGALE)
Brief Title: Study to Assess Functionality, Reliability, and Performance of a Pre-filled Syringe With Benralizumab Administered at Home
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3250C00029
Record Dates: First submitted 2015-03-12; First posted 2015-04-16 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Asthma
Keywords: Asthma,; Bronchial Diseases,; Respiratory Tract Diseases,; Lung Diseases,; Obstructive Lung Diseases,; Benralizumab
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Benralizumab 30 mg (Experimental): Benralizumab administered subcutaneously every 4 weeks
  Interventions: Biological: Benralizumab

INTERVENTIONS:
Biological: Benralizumab — Benralizumab administered subcutaneously every 4 weeks

SUMMARY:
The purpose of the study is to assess functionality, performance, and reliability of an accessorized pre-filled syringe (APFS) with benralizumab administered subcutaneously (SC) in an at-home setting reported by the patient or caregiver, and to confirm the safety and clinical benefit of benralizumab administration in asthma patients with severe asthma.

ELIGIBILITY:
Inclusion criteria

* Written informed consent for study participation must be obtained prior to any study related procedures being performed and according to international guidelines and/or applicable European Union (EU) guidelines
* Male and female patients aged 18 to 75 years of age at the time of Visit 1
* Patient or caregiver must be willing and able to self-administer the IP (Investigational product). Caregiver must be age of consent or older at the time of Visit 1, if applicable
* Weight of ≥40 kg
* Evidence of asthma as documented by either: Airway reversibility (FEV1 ≥12% and 200 ml) demonstrated at Visit 1 or 2 OR documented in the previous 12 months OR; Airflow variability in FEV1 ≥20% between pulmonary function testing documented in the 12 months prior to V2 OR; Airflow variability shown by >20% diurnal variability in peak flow observed in the patient's asthma action plan
* Documented history of current treatment with ICS (Inhaled corticosteroids) and LABA (Long-acting β2 agonists). The ICS and LABA can be parts of a combination product or given by separate inhalers. The ICS dose must be greater than or equal to 500 μg/day fluticasone propionate dry powder formulation or equivalent daily. For ICS/LABA combination preparations, both the mid- and high-strength maintenance doses approved in the local country will meet this ICS criterion. Additional asthma controller medications (e.g., LTRAs (Leukotriene receptor antagonists), tiotropium, theophylline, oral corticosteroids) are allowed
* Morning pre-bronchodilator (pre-BD) FEV1 of >50% predicted at Visit 1 or Visit 2
* Not well controlled asthma as documented by either: An ACQ6 (Asthma Control Questionnaire 6) ≥1.5 OR; A peak flow of 60-80% predicted OR; An exacerbation, one or more, that required oral or systemic corticosteroids in the previous year OR; Any one of the following assessed by patient recall over the previous 2-4 weeks: Asthma symptoms >2 days/week; OR / Nighttime awakenings 1 or more/week; OR / Short acting beta2-agonist use for symptom control (not for prevention of exercise induced asthma) >2 days/week

Exclusion criteria:

* Clinically important pulmonary disease other than asthma (eg, active lung infection, COPD (Chronic obstructive pulmonary disease), bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia) or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (eg, allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome)
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could: Affect the safety of the patient throughout the study; Influence the findings of the studies or their interpretations; Impede the patient's ability to complete the entire duration of study
* Known history of allergy or reaction to the IP formulation
* History of anaphylaxis to any biologic therapy
* History of Guillain-Barré syndrome
* A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy
* Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date informed consent is obtained or during the screening period
* Any clinically significant abnormal findings in physical examination, vital signs, hematology, clinical chemistry, or urinalysis during screening period, which in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2016-03-14 (Actual); Study Completion 2016-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary T. Ferguson, MD, PC, Principal Investigator — Pulmonary Research Institute of Southeast Michigan
Locations (23):
- United States (12):
  - Research Site, Fountain Valley, California
  - Research Site, Walnut Creek, California
  - Research Site, Celebration, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Albany, Georgia
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Bellevue, Nebraska
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, San Antonio, Texas
- Canada (11):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec

REFERENCES:
- [Background] Ferguson GT, Mansur AH, Jacobs JS, Hebert J, Clawson C, Tao W, Wu Y, Goldman M. Assessment of an accessorized pre-filled syringe for home-administered benralizumab in severe asthma. J Asthma Allergy. 2018 Apr 5;11:63-72. doi: 10.2147/JAA.S157762. eCollection 2018. PMID 29670379
- See also: Related Info — http://doi.org/10.2147/JAA.S157762
- See also: Redacted CSP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3529&filename=D3250C00029_Clinical%20Study%20Protocol_GREGALE%20-%20Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 162 participants signed informed consent, 116 participants receive treatment with benralizumab 30 mg at every 4 weeks schedule.
Groups:
- Benra 30 mg: Benralizumab administered subcutaneously every 4 weeks
Period: Overall Study
Arm/Group | Benra 30 mg
Started | 116
Completed | 112
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 52

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Patients/Caregivers Who Successfully Administered Benralizumab 30 mg Subcutaneously (SC) by Injection With an APFS at Home
Description: Number (%) of patients/caregivers who successfully administered benralizumab with an APFS at home among those who have been deemed by the Principal Investigator to be suitable for at-home administration and are still in the study. A successful administration is defined as an injection completed, an answer of "Yes" to all 5 questions in the Functioning Device Return Questionnaire for the GREGALE Clinical Study (Appendix to the Clinical Study Protocol), and adequately passed the visual inspection and function tests. The percentage is calculated among all patients/caregivers who had been deemed by the Principal Investigator to be suitable for at home administration and were still in the study at the time point.
Time Frame: Week 12, Week 16, and Weeks 12 and 16
Population: Full analysis set - all patients who were administered for at least one dose of Benralizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 116
Participants
  Week 12: number analyzed (Participants) | 114
  Week 12 | 112
  Week 16: number analyzed (Participants) | 109
  Week 16 | 108
  Weeks 12 and 16: number analyzed (Participants) | 114
  Weeks 12 and 16 | 106
Statistical Analysis 1: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 12); Percentage = 98.2, 95% CI [93.81 to 99.79] — Percentage of patients who successfully administered benralizumab with an APFS at home (Week 12)
Statistical Analysis 2: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 16); Percentage = 99.1, 95% CI 2-sided [94.99 to 99.98] — Percentage of patients who successfully administered benralizumab with an APFS at home (Week 16)
Statistical Analysis 3: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 12 and 16); Percentage = 93.0, 95% CI 2-sided [86.64 to 96.92] — Percentage of patients who successfully administered benralizumab with an APFS at home (Week 12 and 16)

2. Primary Outcome: Number and Percentage of Returned APFS Used to Administer Benralizumab at Home That Have Been Evaluated as Functional
Description: Number (%) of returned APFS used to administer benralizumab at home that have been evaluated as functional among all returned APFS used to administer benralizumab at home. A functional APFS is defined as an answer of "Yes" to all the questions in the visual inspection and function tests. The percentage is calculated among all returned APFS at the specified time point.
Time Frame: Week 12, Week 16
Population: Full analysis set - all patients who were administered for at least one dose of Benralizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 116
Participants
  Week 12: number analyzed (Participants) | 114
  Week 12 | 113
  Week 16: number analyzed (Participants) | 109
  Week 16 | 108
Statistical Analysis 1: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 12); Percentage = 99.1, 95% CI 2-sided [95.21 to 99.98] — Percentage of patients returned functional APFS administered at home (Week 12)
Statistical Analysis 2: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper Pearson Exact CI; One sample confidence interval (Week 16); Percentage = 99.1, 95% CI 2-sided [94.99 to 99.98] — Percentage of patients returned functional APFS administered at home (Week 16)

3. Primary Outcome: Number and Percentage of APFS Used to Administer Benralizumab at Home or in the Clinic and Have Been Reported as Malfunctioning (Product Complaints)
Description: Number (%) of APFS used to administer benralizumab at home or in the clinic and have been reported as malfunctioning (Product Complaints). The percentage is calculated based on APFS dispensed and used for the specified time point.
Time Frame: Weeks 0, 4, 8, 12, 16, 0 to 8, 12 to 16, and 0 to 16
Population: Number of Units analyzed per row represents number of accessorized pre-filled syringes used at each time point.
Measure: Count of Units; unit: Accessorized Pre-filled Syringe
Units Other Than Participants: Accessorized Pre-filled Syringe
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 116
Number analyzed (Accessorized Pre-filled Syringe) | 573
Accessorized Pre-filled Syringe
  Week 0: number analyzed (Accessorized Pre-filled Syringe) | 116
  Week 0 | 0
  Week 4: number analyzed (Accessorized Pre-filled Syringe) | 117
  Week 4 | 1
  Week 8: number analyzed (Accessorized Pre-filled Syringe) | 115
  Week 8 | 0
  Week 12: number analyzed (Accessorized Pre-filled Syringe) | 116
  Week 12 | 0
  Week 16: number analyzed (Accessorized Pre-filled Syringe) | 109
  Week 16 | 0
  Week 0 to 8: number analyzed (Accessorized Pre-filled Syringe) | 348
  Week 0 to 8 | 1
  Week 12 to 16: number analyzed (Accessorized Pre-filled Syringe) | 225
  Week 12 to 16 | 0
  Week 0 to 16 | 1
Statistical Analysis 1: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 0); Percentage = 0.0, 95% CI 2-sided [0.00 to 3.13] — Percentage of mulfunctioning APFS used to administer benralizumab at home or clinic (Week 0)
Statistical Analysis 2: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 4); Percentage = 0.9, 95% CI 2-sided [0.02 to 4.67] — Percentage of malfunctioning APFS used to administer benralizumab at home or clinic (Week 4)
Statistical Analysis 3: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 8); Percentage = 0.0, 95% CI 2-sided [0.00 to 3.16] — Percentage of malfunctioning APFS used to administer benralizumab at home or clinic (Week 8)
Statistical Analysis 4: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 12); Percentage = 0.0, 95% CI 2-sided [0.00 to 3.13] — Percentage of malfunctioning APFS used to administer benralizumab at home or clinic (Week 12)
Statistical Analysis 5: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-Pearson Exact CI; One sample Confidence Interval (Week 16); Percentage = 0, 95% CI 2-sided [0 to 3.33] — Percentage of malfunctioning APFS used to administer benralizumab at home or clinic (Week 16)
Statistical Analysis 6: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 0 to 8); Percentage = 0.3, 95% CI 2-sided [0.01 to 1.59] — Percentage of malfunctioning APFS used to administer benralizumab at home or clinic (Week 0 to 8)
Statistical Analysis 7: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 12 to 16); Percentage = 0.0, 95% CI 2-sided [0.00 to 1.63] — Percentage of malfunctioning APFS used to administer benralizumab at home or clinic (Week 12 to 16)
Statistical Analysis 8: Comparison: Benra 30 mg; Test type: Superiority or Other; Clopper-pearson Exact CI; One sample Confidence Interval (Week 0 to 16); Percentage = 0.2, 95% CI 2-sided [0.00 to 0.97] — Percentage of malfunctioning APFS used to administer benralizumab at home or clinic (Week 0 to 16)

4. Secondary Outcome: The Effect of Benralizumab on Asthma Control Metrics in Terms of Change From Baseline in Mean Asthma Control Questionnaire-6 (ACQ-6) Score
Description: The effect of benralizumab on asthma control metrics in terms of change from baseline in mean Asthma Control Questionnaire-6 (ACQ-6) score. ACQ-6 score is defined as the average of the first 6 items of the ACQ questionnaire on symptoms, activity limitations, and rescue medication. Baseline is defined as the last non-missing observation prior to the first dose of study treatment. ACQ-6 contains one bronchodilator question and 5 symptom questions. Questions are rated from 0 (totally controlled) to 6 (severely uncontrolled). Mean ACQ-6 score is the average of the responses. Smaller score indicates better controlled asthma.
Time Frame: Week 0 (baseline) and weeks 4, 8, 12, 16, 20
Population: Full analysis set - all patients who were administered for at least one dose of Benralizumab.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 116
Scores on a scale
  Week 4 | -0.53 (0.71)
  Week 8: number analyzed (Participants) | 115
  Week 8 | -0.54 (0.80)
  Week 12: number analyzed (Participants) | 114
  Week 12 | -0.72 (0.86)
  Week 16: number analyzed (Participants) | 109
  Week 16 | -0.82 (0.87)
  Week 20: number analyzed (Participants) | 111
  Week 20 | -0.73 (0.93)

5. Secondary Outcome: The Pharmacokinetics (PK) of Benralizumab in the Terms of PK Parameters: Serum Concentration of Benralizumab
Description: Mean PK Concentration at each visit
Time Frame: Baseline, Week 8, Week 20, and Week 28
Population: PK analysis set - include all patients who had at least one quantifiable serum PK observation post first dose of Benralizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 116
ng/mL
  Baseline: number analyzed (Participants) | 115
  Baseline | NA (NA) — Value is less than lower limit of quantification
  Week 8: number analyzed (Participants) | 113
  Week 8 | 1031.644 (53.547)
  Week 20: number analyzed (Participants) | 111
  Week 20 | 802.197 (267.033)
  Week 28: number analyzed (Participants) | 111
  Week 28 | 56.330 (499.728)

6. Secondary Outcome: The Pharmacodynamics of Benralizumab in the Terms of Peripheral Blood Eosinophil Levels
Description: Blood eosinophil counts by timepoint
Time Frame: Baseline, Week 20, and Week 28
Population: Full analysis set - all patients who were administered for at least one dose of Benralizumab.
Measure: Mean (Standard Deviation); unit: cells/ uL
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 116
cells/ uL
  Baseline | 362.2 (322.01)
  Week 20: number analyzed (Participants) | 110
  Week 20 | 13.0 (56.33)
  Week 28: number analyzed (Participants) | 111
  Week 28 | 47.1 (141.50)

7. Secondary Outcome: The Immunogenicity of Benralizumab in the Terms of Anti-drug Antibodies (ADA)
Description: Anti-drug antibodies (ADA) responses at baseline and post baseline. Persistently positive is defined as positive at >=2 post-baseline assessments (with >=16 weeks between first and last positive) or positive at last post-baseline assessment. Transiently positive is defined as having at least one post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive
Time Frame: Baseline until Week 28
Population: Full analysis set - all patients who were administered for at least one dose of Benralizumab.
Measure: Number; unit: Participants
Arm/Group | Benra 30 mg
Number analyzed (Participants) | 116
Participants
  Positive at any visit | 17
  Base- and Post-baseline Positive | 2
  Only post-baseline positive | 13
  Only baseline positive | 2
  Persistently Positive | 14
  Transiently Positive | 1

ADVERSE EVENTS:
Arm/Group | Benra 30 mg
All-Cause Mortality (participants affected / at risk) | 0/116
Serious Adverse Events (participants affected / at risk) | 7/116
Other Adverse Events (participants affected / at risk) | 43/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=116)
Colitis (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg (N=116)
Bronchitis (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 16 (19)
Sinusitis (Infections and infestations) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 13 (14)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Headache (Nervous system disorders) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.